CLINICAL TRIAL: NCT01237366
Title: A Pilot RCT of Expressive Writing With HIV-Positive Methamphetamine Users
Brief Title: Study Targeting Affect Regulation
Acronym: STAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R03DA029423 (NIH)
Record Dates: First submitted 2010-11-01; First posted 2010-11-09 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: HIV; AIDS; Substance Use Disorders
Keywords: HIV/AIDS; Methamphetamine; Trauma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reslient Affective Processing Therapy (RAPT) (Experimental)
  Interventions: Behavioral: Resilient Affective Processing Therapy (RAPT)
- Attention-Control (No Intervention): Participants will complete 7 sessions where they will be asked to write about neutral topics and complete psychological measures for the purposes of matching for attention and reimbursement.

INTERVENTIONS:
Behavioral: Resilient Affective Processing Therapy (RAPT) — Participants will be asked to complete 7 intervention sessions which include: 1) expressive writing exercises that focus on exploring thoughts and feelings surrounding a difficult life experience; and 2) stress management skills training to assist participants with managing any acute increases in distress that arise following the writing experience.
  Arms: Reslient Affective Processing Therapy (RAPT)

SUMMARY:
This Phase Ib pilot RCT will examine the safety, feasibility, and acceptability of a multi-component intervention to address traumatic stress symptoms among HIV-positive, methamphetamine-using men who have sex with men (MSM). Following a baseline assessment, 56 participants will be randomized to receive either: 1) a 7-session intervention to address traumatic stress related to living with HIV/AIDS; or 2) a 7-session, attention-control condition. Follow-up assessments will be administered at 1 and 3 months post-randomization.

DETAILED DESCRIPTION:
In the multi-component intervention protocol, participants will complete expressive writing exercises where they will be asked to write about difficult life experiences. Following expressive writing, participants will receive stress management skills training to assist them with managing any acute increases in distress that arise from the writing experience. Participants in the attention-control condition will write about neutral topics and complete psychological measures. The overarching goals of this Phase Ib RCT will be to: 1) examine the feasibility and acceptability of the intervention and attention-control; and 2) determine whether intervention participants report reductions in traumatic stress symptoms over the 3 months following randomization. Findings from this Phase Ib trial will inform our efforts to implement a more definitive RCT of this intervention with HIV-positive, methamphetamine-using MSM.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak English
* Self-identify as a man who has sex with men
* Have been diagnosed with HIV for at least 3 months
* Provide evidence of HIV-positive serostatus
* Report using methamphetamine during the past 30 days

Exclusion Criteria:

* Do not have the capacity to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Traumatic stress symptom severity | 3-month follow-up
  Our team will use the Impact of Event Scale to measure the self-reported severity of traumatic stress symptoms related to HIV/AIDS.

SECONDARY OUTCOMES:
Psychological reactivity to expressive writing | 1-month follow-up
  Participants will complete measures of subjective distress and craving of stimulants (i.e., methamphetamine, cocaine, and crack) before and after each expressive writing exercise to provide an index of habituation. Habituation is defined as a 50% reduction in the psychological reactivity to the expressive writing experience using these self-report measures.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Carrico, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for AIDS Prevention Studies, San Francisco, California, United States